CLINICAL TRIAL: NCT04315714
Title: Impact of a Yoga Intervention on Chronic Abdominal Pain, and Associations With the Metagenome and Metabolome in Participants With IBS
Brief Title: Impact of a Yoga Intervention on Pain and Multiomics in Participants With IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kristen Weaver, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00089815; 1P30NR016579-01 (NIH)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain
Keywords: Irritable bowel syndrome; IBS; Yoga; Microbiome; Abdominal pain; Metagenome; Metabolome
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: This will be a randomized, controlled trial crossover design, evaluating a yoga intervention, delivered online/virtually via Zoom, with a wait-list control condition for 6 weeks. Study participants will be crossed over to the alternative intervention for an additional 6 weeks, with total intervention time of 12 weeks. Twenty participants with irritable bowel syndrome (IBS) and 20 healthy controls (HC) will be recruited; 10 participants with IBS will be randomized to the yoga intervention at the beginning of the trial, and 10 participants with IBS randomized to the waitlist control condition. Likewise, 10 HC participants will be randomized to the yoga intervention at the beginning of the trial, and 10 HC will be randomized to the waitlist control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IBS Yoga Intervention (delivered online/virtually via Zoom) (Experimental): Ten participants with IBS will be randomized to the 6-week yoga intervention at the beginning of the trial, followed by the 6-week control condition (observation/active monitoring).
  Interventions: Other: Yoga Program
- IBS Waitlist Control Condition (Experimental): Ten participants with IBS will be randomized to the 6-week waitlist control condition (observation/active monitoring) at the beginning of the trial, followed by the 6-week yoga intervention.
  Interventions: Other: Yoga Program
- HC Yoga Intervention (delivered online/virtually via Zoom) (Experimental): Ten participants serving as HC will be randomized to the 6-week yoga intervention at the beginning of the trial, followed by the 6-week control condition (observation/active monitoring).
  Interventions: Other: Yoga Program
- HC Waitlist Control Condition (Experimental): Ten participants serving as HC will be randomized to the 6-week waitlist control condition (observation/active monitoring) at the beginning of the trial, followed by the 6-week yoga intervention.
  Interventions: Other: Yoga Program

INTERVENTIONS:
Other: Yoga Program — Six-week, twice weekly, 60-minute private yoga program (delivered online/virtually via Zoom).

SUMMARY:
The purpose of this research study is to see if a six-week yoga program delivered online/virtually via Zoom, reduces abdominal pain in people with irritable bowel syndrome (IBS). This study also looks at whether the yoga program changes the composition of microorganisms in the gut and their metabolites, and compares the program in people with IBS versus healthy people (also known as "healthy controls" or "HC"). People in this study are randomized (like flipping a coin) to one of two conditions: half of the people attend the online/virtual private yoga program delivered via Zoom for the first six-weeks, and half of the people wait for six-weeks and then attend the online/virtual private yoga program for six-weeks. The hypothesis of this study is that the practice of yoga induces shifts in the gut microbiota and microbial-derived metabolites, which will correlate with diminished abdominal pain.

DETAILED DESCRIPTION:
Chronic abdominal pain is a hallmark feature of irritable bowel syndrome (IBS)1; a prevalent2, costly disorder3 that disproportionately affects the female sex4. IBS is often comorbid with psychiatric disorders and other pain-related conditions, and although pathophysiology is not yet fully understood, alterations in the gut microbiota, epithelial barrier and immune response are among factors noted to play a role5. Bidirectional signaling between the brain, the gut, and its microbiome is relevant to the disorder of IBS, with top-down signaling including through the autonomic nervous system, and bottom-up signaling through microbial-derived intermediates including secondary bile acids, short-chain fatty acids (SCFA), and tryptophan metabolites6. Diet and lifestyle are critical determinants of the microbiota composition7, thus interventions which modulate the microbiota and affect microbial-derived intermediates, have the potential to improve patient symptomatology. A recent meta-analysis of common dietary interventions for IBS, however, demonstrates insufficient evidence to recommend a gluten-free diet, and very low quality evidence supporting the efficacy a low fermentable oligo-di-and monosaccharides and polyols (FODMAP) diet to reduce symptoms of IBS8. Therefore, a need exists to identify alternative lifestyle interventions for patients with IBS, and given the acknowledged role of the microbiota in pathophysiology, enhance our understanding of how such interventions modulate the microbiota, affect microbial-derived intermediates, and influence patient symptoms of chronic abdominal pain.

A lifestyle intervention of increasing interest in IBS research is physical activity; a recent systematic review suggests exercise to improve gastrointestinal (GI) symptoms, anxiety, depression, stress, and quality of life9. The practice of yoga, in particular, benefits anxiety, quality of life and GI symptoms in patients with IBS10, although physiological underpinnings of this effect remain understudied in IBS. A recent meta-analysis of randomized controlled trials comparing the practice of yoga asanas (body postures) with active controls across patient populations, reports yoga to improve cortisol, cytokines, autonomic measures, fasting blood glucose and lipids11. An additional pathway by which yoga may affect symptomatology in IBS is along the gut microbiota-skeletal muscle axis. Preclinical findings report the gut microbiota to influence skeletal muscle mass and function in mice, with germ free mice displaying altered amino acid metabolism12. Importantly, this gut-muscle axis appears bi-directional, in that microbiota may modulate muscle function through nutrient synthesis and biotransformation, whereas regular exercise can modulate the composition of the microbiota, and enhance gut microbiota diversity13. Exercise training has been found to increase concentrations of SCFA including butyrate14, a microbial end product with beneficial effects upon intestinal inflammation, immunity and gut barrier function15, and levels of which have been noted as altered in patients with IBS in comparison with healthy controls (HC)16. The gut microbiota of patients with IBS compared with HC, consistently includes lower microbial α-diversity, decreased levels of Bacteroidetes, increased levels of Firmicutes, and increased F/B ratio17. Metagenomics and metabolomics used in combination, can provide a comprehensive overview of microbiome-host interactions18. This was demonstrated by a recent investigation of children with IBS and HC, in which IBS children were found to be enriched in bacterial taxa (e.g. Flavonifractor plautii), metagenomics functional profile (e.g. amino acid metabolism), higher-order metabolites (e.g. secondary bile acids), and associations were noted with abdominal pain19.

The investigators of this study hypothesize that participants with IBS differ from HC in lower microbial α-diversity and reduced SCFA (specifically butyrate), which will be associated with abdominal pain. Furthermore, the investigators of this study hypothesize that the practice of yoga induces shifts in the gut microbiota and microbial-derived metabolites, specifically butyrate, which will correlate with diminished abdominal pain. To test these hypotheses, the investigators of this study propose the following two aims:

Specific Aim 1: Identify differences in microbial features and metabolites among participants with IBS and HC at baseline, and evaluate associations with participant characteristics

Specific Aim 2: Determine if a 6-week yoga intervention delivered online/virtually via Zoom, reduces abdominal pain among participants with IBS, and evaluate associations with microbial features and metabolites.

Findings from this study will enhance our understanding of the interplay between the microbiota, microbial-derived intermediates and pain in patients with IBS. Furthermore, this research will facilitate the identification of relevant microbial features and metabolites that may prove modifiable, and work towards diminishing the public health burden surrounding chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read/write in English
* Access to smartphone/computer/email; Internet and camera access for online/virtual yoga sessions via Zoom
* Physical ability to engage in twice weekly yoga for 6 weeks (60 minutes each session), with physical clearance provided by current healthcare provider
* Diagnosis of IBS and IBS subtype (for cases), with documentation provided by current healthcare provider
* Self-report average, abdominal pain over past 7 days ≥ 3 (for cases: on 0-10 scale)
* Willingness to participate in all study procedures

Exclusion Criteria:

* Regular yoga practice (past 3 months)
* Recent antibiotic use (past 3 months)
* Consumption of a strict vegan/vegetarian diet
* Plan to initiate prebiotic/synbiotic/probiotic use during study period
* Any medical condition (cardiac, pulmonary, neurological, musculoskeletal, immunological etc.) that would preclude engagement in the yoga intervention
* Any organic gastrointestinal condition (inflammatory bowel disease: Crohn's disease, Ulcerative Colitis, active H. pylori infection, etc.)
* Severe comorbid pain or psychiatric condition requiring recent hospitalization
* Pregnancy, or plans to become pregnant during study period
* Unwilling to participate in study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Changes in Abdominal Pain | 6 weeks
  To test the hypothesis that a 6-week yoga intervention, delivered online/virtually via Zoom, reduces abdominal pain among participants with IBS. Participants will be asked to rate their average level of abdominal pain over the past 7 days on a 0-10 scale, where 0 represents no pain, and 10 represents the worst imaginable pain.

SECONDARY OUTCOMES:
Baseline Metagenomics | Baseline
  To identify baseline differences between participants with IBS and HC in the gut microbiota, its genome, and potential functions; evaluated through the collection of stool samples.
Baseline Metabolomics | Baseline
  To identify baseline differences between participants with IBS and HC in metabolites; analyzed through the collection of stool samples.
Changes in Metagenomics | 6 weeks
  To test the hypothesis that a 6-week yoga intervention induces changes to the metagenome among participants with IBS and HC; evaluated through the collection of stool samples.
Changes in Metabolomics | 6 weeks
  To test the hypothesis that a 6-week yoga intervention induces changes to the metabolome among participants with IBS and HC; analyzed through the collection of stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen R Weaver, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The funder of this study, the National Institute of Nursing Research (NINR), National Institutes of Health (NIH), requires that individual participant data be de-identified, and shared in a data repository, the Biomedical Research Informatics Computing System (BRICS). Participants will be assigned an NIH Global Unique Identifier (GUID), under which the following data will be shared: age, gender, race, ethnicity, education level, caregiver status, employment status, marital or partner status, and household member total count. In addition, questionnaire responses pertaining to the following symptoms will be shared in BRICS via the GUID: anxiety, depression, constipation, diarrhea, global health, pain and sleep. To create a GUID for each participant, the following information will be collected, but will not be shared in the data repository: participants' name at birth, city and country of birth.
Time Frame: Data will be shared one year after the project end date and stored indefinitely, unless the participant requests that their data be removed.
Access Criteria: Requests to access data from BRICS are reviewed and approved by the NINR/BRICS Operations team. Steps to request access include reading and submitting a signed BRICS data use certification (DUC), and submitting an Informatics System Access Request (ISAR). Protecting data privacy, security and confidentiality are among expectations of the BRICS policy for requesting data access.
URL: http://cdrns.nih.gov/

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part I: overall and upper gastrointestinal diseases. Gastroenterology. 2009 Feb;136(2):376-86. doi: 10.1053/j.gastro.2008.12.015. Epub 2009 Jan 3. No abstract available. PMID 19124023
- [Background] Sperber AD, Dumitrascu D, Fukudo S, Gerson C, Ghoshal UC, Gwee KA, Hungin APS, Kang JY, Minhu C, Schmulson M, Bolotin A, Friger M, Freud T, Whitehead W. The global prevalence of IBS in adults remains elusive due to the heterogeneity of studies: a Rome Foundation working team literature review. Gut. 2017 Jun;66(6):1075-1082. doi: 10.1136/gutjnl-2015-311240. Epub 2016 Jan 27. PMID 26818616
- [Background] Enck P, Aziz Q, Barbara G, Farmer AD, Fukudo S, Mayer EA, Niesler B, Quigley EM, Rajilic-Stojanovic M, Schemann M, Schwille-Kiuntke J, Simren M, Zipfel S, Spiller RC. Irritable bowel syndrome. Nat Rev Dis Primers. 2016 Mar 24;2:16014. doi: 10.1038/nrdp.2016.14. PMID 27159638
- [Background] Osadchiy V, Martin CR, Mayer EA. The Gut-Brain Axis and the Microbiome: Mechanisms and Clinical Implications. Clin Gastroenterol Hepatol. 2019 Jan;17(2):322-332. doi: 10.1016/j.cgh.2018.10.002. Epub 2018 Oct 4. PMID 30292888
- [Background] Barbara G, Feinle-Bisset C, Ghoshal UC, Quigley EM, Santos J, Vanner S, Vergnolle N, Zoetendal EG. The Intestinal Microenvironment and Functional Gastrointestinal Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00219-5. doi: 10.1053/j.gastro.2016.02.028. Online ahead of print. PMID 27144620
- [Background] Dionne J, Ford AC, Yuan Y, Chey WD, Lacy BE, Saito YA, Quigley EMM, Moayyedi P. A Systematic Review and Meta-Analysis Evaluating the Efficacy of a Gluten-Free Diet and a Low FODMAPs Diet in Treating Symptoms of Irritable Bowel Syndrome. Am J Gastroenterol. 2018 Sep;113(9):1290-1300. doi: 10.1038/s41395-018-0195-4. Epub 2018 Jul 26. PMID 30046155
- [Background] Zhou C, Zhao E, Li Y, Jia Y, Li F. Exercise therapy of patients with irritable bowel syndrome: A systematic review of randomized controlled trials. Neurogastroenterol Motil. 2019 Feb;31(2):e13461. doi: 10.1111/nmo.13461. Epub 2018 Sep 19. PMID 30232834
- [Background] Schumann D, Anheyer D, Lauche R, Dobos G, Langhorst J, Cramer H. Effect of Yoga in the Therapy of Irritable Bowel Syndrome: A Systematic Review. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1720-1731. doi: 10.1016/j.cgh.2016.04.026. Epub 2016 Apr 22. PMID 27112106
- [Background] Pascoe MC, Thompson DR, Ski CF. Yoga, mindfulness-based stress reduction and stress-related physiological measures: A meta-analysis. Psychoneuroendocrinology. 2017 Dec;86:152-168. doi: 10.1016/j.psyneuen.2017.08.008. Epub 2017 Aug 30. PMID 28963884
- [Background] Lahiri S, Kim H, Garcia-Perez I, Reza MM, Martin KA, Kundu P, Cox LM, Selkrig J, Posma JM, Zhang H, Padmanabhan P, Moret C, Gulyas B, Blaser MJ, Auwerx J, Holmes E, Nicholson J, Wahli W, Pettersson S. The gut microbiota influences skeletal muscle mass and function in mice. Sci Transl Med. 2019 Jul 24;11(502):eaan5662. doi: 10.1126/scitranslmed.aan5662. PMID 31341063
- [Background] Ticinesi A, Lauretani F, Tana C, Nouvenne A, Ridolo E, Meschi T. Exercise and immune system as modulators of intestinal microbiome: implications for the gut-muscle axis hypothesis. Exerc Immunol Rev. 2019;25:84-95. PMID 30753131
- [Background] Allen JM, Mailing LJ, Niemiro GM, Moore R, Cook MD, White BA, Holscher HD, Woods JA. Exercise Alters Gut Microbiota Composition and Function in Lean and Obese Humans. Med Sci Sports Exerc. 2018 Apr;50(4):747-757. doi: 10.1249/MSS.0000000000001495. PMID 29166320
- [Background] Riviere A, Selak M, Lantin D, Leroy F, De Vuyst L. Bifidobacteria and Butyrate-Producing Colon Bacteria: Importance and Strategies for Their Stimulation in the Human Gut. Front Microbiol. 2016 Jun 28;7:979. doi: 10.3389/fmicb.2016.00979. eCollection 2016. PMID 27446020
- [Background] Sun Q, Jia Q, Song L, Duan L. Alterations in fecal short-chain fatty acids in patients with irritable bowel syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Feb;98(7):e14513. doi: 10.1097/MD.0000000000014513. PMID 30762787
- [Background] Duan R, Zhu S, Wang B, Duan L. Alterations of Gut Microbiota in Patients With Irritable Bowel Syndrome Based on 16S rRNA-Targeted Sequencing: A Systematic Review. Clin Transl Gastroenterol. 2019 Feb;10(2):e00012. doi: 10.14309/ctg.0000000000000012. PMID 30829919
- [Background] Mayneris-Perxachs J, Fernandez-Real JM. Exploration of the microbiota and metabolites within body fluids could pinpoint novel disease mechanisms. FEBS J. 2020 Mar;287(5):856-865. doi: 10.1111/febs.15130. Epub 2019 Nov 24. PMID 31709683
- [Background] Hollister EB, Oezguen N, Chumpitazi BP, Luna RA, Weidler EM, Rubio-Gonzales M, Dahdouli M, Cope JL, Mistretta TA, Raza S, Metcalf GA, Muzny DM, Gibbs RA, Petrosino JF, Heitkemper M, Savidge TC, Shulman RJ, Versalovic J. Leveraging Human Microbiome Features to Diagnose and Stratify Children with Irritable Bowel Syndrome. J Mol Diagn. 2019 May;21(3):449-461. doi: 10.1016/j.jmoldx.2019.01.006. Epub 2019 Apr 17. PMID 31005411